CLINICAL TRIAL: NCT01582971
Title: Home-Based Symptom Management Via Reflexology for Breast Cancer Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Michigan State University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Gwen Wyatt, Professor, Michigan State University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1R01CA157459-01 (NIH); 1R01CA157459-01 (NIH)
Record Dates: First submitted 2012-04-17; First posted 2012-04-23 (Estimated); Results first posted 2017-10-02 (Actual); Last update posted 2018-04-18 (Actual); Status verified 2018-03

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Reflexology; Complementary
MeSH Terms: conditions — Breast Neoplasms | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Intervention (Experimental): Reflexology: 4 weekly foot reflexology sessions delivered by friend/family member
  Interventions: Other: Reflexology
- Control (No Intervention): Standard medical care: no reflexology

INTERVENTIONS:
Other: Reflexology — Friend/family member trained in foot reflexology protocol by certified reflexologist; friend/family member provides 4 weekly sessions to patient
  Arms: Intervention

SUMMARY:
The purpose of this project is to test foot reflexology delivered by a friend or family member in the home for women with breast cancer. The primary aims of the proposed study in a sample of women with breast cancer receiving chemotherapy and/or hormonal therapy are to determine the effects of 4 family- or friend-delivered weekly reflexology sessions compared to an attention control group.

DETAILED DESCRIPTION:
This project tests the benefits of a home-based intervention of foot reflexology for improving health-related quality of life (HRQOL) including symptom responses, functioning, and health perceptions in women treated with chemotherapy for advanced breast cancer. Reflexology applies a firm walking-motion during sessions and is based on the premise that the foot has reflexes mirroring organs of the body. Symptom burden is the strongest predictor of HRQOL for cancer patients. This project brings together expertise from nursing, reflexology, communication, statistics, and health economics. The primary specific aims, in a sample of women with advanced breast cancer receiving chemotherapy, are to determine the effects of a 4-week, home-based reflexology intervention delivered by a friend/family provider compared to attention control for improvement of:

1. HRQOL including symptoms, functioning, and health perception at study weeks 5 and 11.

   The investigators hypothesize that the reflexology group will have better HRQOL (symptoms, functioning, and health perception) than the attention control group at study weeks 5 and 11.
2. Multiple symptom responses and times-to-response as determined by weekly symptom assessments during the 4-week intervention time.

   The investigators hypothesize that the reflexology group will have a higher proportion of symptoms that respond to the intervention and shorter time-to-symptom-responses than the attention control group.
3. Symptom-related use of unscheduled health services during the 11-week study. The investigators hypothesize that fewer unscheduled services will be used for symptom management over the 11-week study period by women receiving reflexology compared to women in the attention control.

The exploratory aims are to: 1) Explore differences between trial arms in perceptions of social support due to the family- or friend-delivered reflexology sessions at study weeks 5 and 11; 2) Determine if effects of the reflexology intervention on HRQOL are mediated by social support; and 3) Use the newly developed NIH PROMIS standardized symptom and functioning instruments to assess the effects of the reflexology intervention and to compare the responsiveness of PROMIS instruments and existing instruments designed to measure similar constructs.

This project has immense potential to make an effective symptom management intervention accessible to patients in their homes via a friend or family home provider. The investigators will not only intervene to enhance HRQOL but also to evaluate social support and costs associated with unscheduled health services. Effective symptom management provides time and cost savings to clinicians, advances the current state-of-the-science, and promotes adherence to medical treatment that may ultimately enhance survival.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 21
* Diagnosis of breast cancer, Stage III, IV, or Stage I or II with metastasis or recurrence
* Able to perform basic ADLs
* Undergoing chemotherapy and/or hormonal therapy for breast cancer
* Able to speak and understand English
* Have access to a telephone
* Able to hear normal conversation
* Cognitively oriented to time, place, and person (determined via nurse recruiter)

Exclusion Criteria:

* Diagnosis of major mental illness on the medical record and verified by the recruiter
* Residing in a nursing home
* Bedridden
* Currently receiving regular reflexology
* Diagnosis of symptoms of deep vein thrombosis or painful foot neuropathy, which will require medical approval

Min Age: 21 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2012-04-17; Primary Completion 2016-05-01 (Actual); Study Completion 2016-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gwen Wyatt, PhD, RN, Principal Investigator — Michigan State University
Locations (9):
- United States (9):
  - Northwestern, Chicago, Illinois
  - Hurley Medical Center, Flint, Michigan
  - Lemmon-Holton Cancer Center, Grand Rapids, Michigan
  - Breslin Cancer Center, Lansing, Michigan
  - Sparrow Cancer Center, Lansing, Michigan
  - McLaren Macomb, Mount Clemens, Michigan
  - St. Joseph Mercy Oakland Hospital, Pontiac, Michigan
  - Beaumont Hospital, Royal Oak, Michigan
  - St. Johns Providence, Warren, Michigan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sikorskii A, Niyogi PG, Victorson D, Tamkus D, Wyatt G. Symptom response analysis of a randomized controlled trial of reflexology for symptom management among women with advanced breast cancer. Support Care Cancer. 2020 Mar;28(3):1395-1404. doi: 10.1007/s00520-019-04959-y. Epub 2019 Jul 2. PMID 31267277
- [Derived] Luo Z, Wang L, Sikorskii A, Wyatt G. Healthcare service utilization and work-related productivity in reflexology intervention for advanced breast cancer women. Support Care Cancer. 2019 Aug;27(8):2837-2847. doi: 10.1007/s00520-018-4592-4. Epub 2018 Dec 14. PMID 30552595

RESULTS

PARTICIPANT FLOW:
Groups:
- Intervention: Reflexology: 4 weekly foot reflexology sessions delivered by friend/family member.
  Friend/family member was trained in foot reflexology protocol by certified reflexologist.
  Friend/family member provides 4 weekly sessions to patient.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 128 | 128
Completed | 89 | 91
Not Completed | 39 | 37
Not completed — Death | 2 | 1
Not completed — Lost to Follow-up | 18 | 21
Not completed — Withdrawal by Subject | 4 | 2
Not completed — Other | 15 | 13

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 128 | 128 | 256
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.09 (11.62) | 54.80 (10.30) | 56.44 (11.08)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 128 | 128 | 256
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 6 | 11
  Not Hispanic or Latino | 123 | 122 | 245
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 13 | 13 | 26
  White | 105 | 107 | 212
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 10 | 8 | 18
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 128 | 128 | 256

OUTCOME MEASURES:

1. Primary Outcome: The M.D. Anderson Symptom Inventory (MDASI)
Description: The M.D. Anderson Symptom Inventory (MDASI) evaluates severity of 13 symptoms experienced by cancer patients (pain, fatigue, nausea, disturbed sleep, distress, shortness of breath, difficulty remembering, decreased appetite, drowsiness, dry mouth, sadness, vomiting, numbness/tingling) on the scale from 0=symptom not present to 10=as bad as you can imagine. Summed symptom severity score ranging from 0 to 130 was derived. MDASI also assesses how much symptoms interfered with 6 aspects of daily life: general activity, mood, work (including work around the house), relations with other people, walking, and enjoyment of life on the scale from 0=did not interfere to 10=interfered completely. Summed interference score ranging from 0 to 60 was derived.
  Higher symptom severity and interference scores represent worse outcome.
Time Frame: Week 5 and week 11
Population: Patient outcome data collected at week 5 and week 11
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Groups:
- Week 5 Intervention Group; Week 11 Intervention Group: Reflexology: 4 weekly foot reflexology sessions delivered by friend/family member.
  Friend/family member was trained in foot reflexology protocol by certified reflexologist.
  Friend/family member provides 4 weekly sessions to patient.
- Week 5 Control Group; Week 11 Control Group: Standard medical care: no reflexology
Arm/Group | Week 5 Intervention Group | Week 5 Control Group | Week 11 Intervention Group | Week 11 Control Group
Number analyzed (Participants) | 89 | 91 | 89 | 91
units on a scale
  MDASI summed symptom severity | 23.55 (1.52) | 29.69 (1.48) | 26.28 (1.54) | 28.67 (1.52)
  MDASI summed symptom interference | 11.19 (1.16) | 16.04 (1.12) | 12.43 (1.17) | 14.88 (1.16)

2. Primary Outcome: Patient Reported Outcomes Measurement Information System (PROMIS) V 1.0
Description: 1. PROMIS-Physical functioning subscale contains four items. Score for each item ranging from 1 to 5, yielding a total score ranges from 4 to 20. Raw score is converted to a T-score using PROMIS scoring rules. The T-scores have mean 50 and standard deviation 10 for the general population.
  2. PROMIS-Satisfaction with participation in social roles subscale contains four items. Score for each item ranges from 0 to 4, yielding a total score ranges from 0 to 16. Raw score is converted to a T-score using PROMIS scoring rules. The T-scores have mean 50 and standard deviation 10 for the general population.
  Higher scores representing better outcomes in each subscale.
Time Frame: Week 5 and week 11
Population: Participant outcome data collected at week 5 and week 11
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Week 5 Intervention Group | Week 5 Control Group | Week 11 Intervention Group | Week 11 Control Group
Number analyzed (Participants) | 89 | 91 | 89 | 91
units on a scale
  PROMIS-Physical function subscale | 42.06 (0.57) | 41.81 (0.55) | 42.93 (0.57) | 42.80 (0.56)
  PROMIS-Social role subscale | 47.59 (0.78) | 46.86 (0.75) | 48.58 (0.79) | 45.92 (0.78)

3. Primary Outcome: Quality of Life Index (QLI)
Description: The QLI assesses perceived quality of life including health and functioning domain, psychological/spiritual domain, social and economic domain, and family domain. The QLI consists of two sections: one measures respondent's satisfaction with the various domain of life and the other measures the importance of those domains. The satisfaction scores are centered and weighed by the importance scores to obtain the QLI composite score that ranges from 0 to 30 with higher scores representing better outcomes.
Time Frame: Week 5 and week 11
Population: Participant outcome data collected at week 5 and week 11
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Week 5 Intervention Group | Week 5 Control Group | Week 11 Intervention Group | Week 11 Control Group
Number analyzed (Participants) | 89 | 91 | 89 | 91
units on a scale | 22.53 (0.29) | 21.94 (0.28) | 22.69 (0.29) | 22.08 (0.29)

4. Primary Outcome: Use of Unscheduled Health Service
Description: Measured by Conventional Health Service and Productivity Costs to assess the number of unscheduled times the patient visits an emergency room, urgent care center, and hospitalization.
Time Frame: Week 11
Population: Participant outcome data collected at week 11
Measure: Mean (Standard Deviation); unit: unscheduled visits
Arm/Group | Intervention | Control
Number analyzed (Participants) | 89 | 91
unscheduled visits
  Number of emergency room visits | 0.27 (0.78) | 0.65 (2.85)
  Number of urgent care center visits | 0.09 (0.33) | 0.12 (0.39)
  Number of Hospitalizations | 0.76 (1.19) | 1.05 (0.61)

ADVERSE EVENTS:
Time Frame: Adverse events were tracked for unexpected foot effect at weeks 1-11
Description: Adverse events were tracked from patient's report of the unexpected foot effect (UFE) which adapted from the Patient-Reported Outcomes version of Common Terminology Criteria for Adverse Events (PRO-CTCAE) including discomfort, numbness or tingling, discoloration or bruising.
Arm/Group | Intervention | Control
All-Cause Mortality (participants affected / at risk) | 2/128 | 1/128
Serious Adverse Events (participants affected / at risk) | 0/128 | 0/128
Other Adverse Events (participants affected / at risk) | 0/128 | 0/128

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No